CLINICAL TRIAL: NCT00034658
Title: Open Label, Treatment Protocol for the Safety and Efficacy of Posaconazole (SCH 56592) in the Treatment of Invasive Fungal Infections
Brief Title: Open Label Study of Posaconazole in the Treatment of Invasive Fungal Infections (Study P00041)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00041
Record Dates: First submitted 2002-05-01; First posted 2002-05-02 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Mycoses
Keywords: Aspergillosis, Candidiasis, Cryptococcosis,
MeSH Terms: conditions — Mycoses; Aspergillosis; Candidiasis; Cryptococcosis | interventions — posaconazole

INTERVENTIONS:
Drug: Posaconazole

SUMMARY:
This study is designed to evaluate the safety, tolerance and efficacy of Posaconazole (SCH 56592) under an open label, treatment protocol for subjects with invasive fungal infections:

A: which are refractory or resistant to standard antifungal therapies; B: for which there are currently no effective therapies; C: with a prior history of serious, severe or life-threatening toxicities while receiving antifungal therapy; D: with pre-existing organ dysfunction which precludes the administration of standard antifungal therapies.

DETAILED DESCRIPTION:
The current clinical trial is designed to provide posaconazole (SCH 56592) to subjects with invasive fungal infections a)which are refractory or resistant to standard antifungal therapies or b) for which there are currently no effective therapies. Subjects with such invasive fungal infections cannot be enrolled in controlled, randomized clinical trials. Secondly, this clinical trial is also designed to provide posaconazole (SCH 56592) to subjects with invasive fungal infections who c) have experienced serious or severe toxicities while receiving standard antifungal therapies or d) have pre-existing organ dysfunction such as renal dysfunction who require standard antifungal therapy which is precluded because of the toxicities associated with such therapy. This clinical trial also serves to allow collection of preliminary data regarding the safety and efficacy of posaconazole (SCH 56592) against a variety of invasive fungal infections which although serious and life-threatening are sufficiently rare so that they cannot be studied in a controlled, randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria

* Proven or probable invasive fungal infections according to EORTC/MSG criteria.
* IFI are documented to be refractory to standard antifungal therapy OR intolerant to standard therapy.
* Able to take oral medication or take medication via enteral feeding tube.

Exclusion Criteria

* Concurrent progressive neurological disease (except if due to invasive fungal infection)
* Use of medications that are known to interact with azoles and that may lead to life-threatening side to effects.
* Prior enrollment in this study.
* Subjects with a life expectancy of less than 72 hours.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 1998-12; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

REFERENCES:
- [Result] Alexander BD, Perfect JR, Daly JS, Restrepo A, Tobon AM, Patino H, Hardalo CJ, Graybill JR. Posaconazole as salvage therapy in patients with invasive fungal infections after solid organ transplant. Transplantation. 2008 Sep 27;86(6):791-6. doi: 10.1097/TP.0b013e3181837585. PMID 18813103
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html